CLINICAL TRIAL: NCT02098980
Title: Nutritional Intervention of Type II Diabetes Mellitus by Vitamin D in Qatar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Supreme Council Of Health, Qatar (Other Government)
Responsible Party: Principal Investigator, Mohamed Al Thani, Doctor, Supreme Council Of Health, Qatar
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: INDDIQAT Trial; Vitamin D and Diabetes (Other Grant/Funding Number: Qatar National Research Fund/ NPRP No.: 6-273-3-067)
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Vitamin D (Active Comparator): Vitamin D supplement 4000 IU/day for 6 months
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo for 6 months
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Other Names: Placebo

SUMMARY:
There is an association between elevated Type II Diabetes Mellitus (T2DM) risk and low serum levels of vitamin D. It is important to examine whether Vitamin D can enhance oral glucose tolerance in individuals at risk for developing T2DM. As such, the hypothesis suggested is that Vitamin D supplementation (4,000 IU/day) for 24 weeks in pre-diabetic individuals will decrease insulin resistance and the associated metabolic indices linked to the later development of T2DM.

DETAILED DESCRIPTION:
Epidemiologically, there is an association between elevated T2DM risk and low serum levels of vitamin D and suggest that it may protect against the diseases through the improvement of insulin sensitivity as well as secretion and reducing chronic inflammation. Although some of these effects were shown in clinical studies, no study permitted the inference that vitamin D can reduce blood glucose and attenuate inflammation. Post-prandial glucose is the most sensitive to alterations in insulin sensitivity. Therefore, it is rational to examine whether vitamin D can enhance oral glucose tolerance in individuals at risk for developing T2DM and to elucidate the mechanism by which this occurs, i.e. via improved insulin sensitivity or improved insulin secretion, or both. Furthermore, identifying a distinct proteomics-based signature that can be used to distinguish responders to supplementation from non-responders is critical to define the bases for inter-individual variation in response and the effect of vitamin D on the prevention of T2DM. Identification of this proteomics-based signature will enable us to tailor alternative preventive measures to adjust the vitamin D dose to non-responders, leading to more effective and precise intervention protocols.

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant, non-lactating females, aged 18-75
* volunteered to participate by signing the consent form
* BMI ˂ 40kg/ m2
* serum 25(OH) vitamin D3 (25(OH)D) concentration ˂75nmol/L
* fasting serum glucose <7.0 mmol/L
* HOMA insulin resistance index ≥1.3
* presence of any ONE OR MORE of the following risk factors for type 2 diabetes:

  * high BMI (>23)
  * high waist circumference according to IDF ethnic specific values for non- Caucasian (females >80cm; males >90cm)
  * family history of diabetes in first-degree relative (parent or sibling)
  * previous history of gestational diabetes
  * history of high blood glucose, high triglycerides and/or low HDL cholesterol

Exclusion Criteria:

* fasting serum glucose ≥7.0mmol/L
* history of renal failure or liver disease
* serum urea or creatinine >1.8 times upper limit of normal (ULN)
* serum aspartate or alanine transaminase (AST,ALT) >1.5 times ULN
* current use of drug or drugs to treat diabetes or which influence glucose metabolism
* medical or surgical event requiring hospitalization within 3 months of randomization
* presence of any condition affecting nutrient absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Thani, Ph.D., Principal Investigator — Supreme Council of Health
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Al Thani M, Sadoun E, Sofroniou A, Jayyousi A, Baagar KAM, Al Hammaq A, Vinodson B, Akram H, Bhatti ZS, Nasser HS, Leventakou V. The effect of vitamin D supplementation on the glycemic control of pre-diabetic Qatari patients in a randomized control trial. BMC Nutr. 2019 Oct 10;5:46. doi: 10.1186/s40795-019-0311-x. eCollection 2019. PMID 32153959